CLINICAL TRIAL: NCT03079427
Title: Randomized Phase 2 Study of Capecitabine vs Gemcistabine Plus Cisplatin in Patients With Resected Extrahepatic Cholangiocarcinoma With Regional Lymph Node Metastasis
Brief Title: Adjuvant Capecitabine vs Gemcitabine Plus Cisplatin in Resected Extrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bundang CHA Hospital (Other); Seoul St. Mary's Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Baek-Yeol Ryoo, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asan-ONCHBP-2017-001
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Cholangiocarcinoma; Biliary Tract Cancer; Adjuvant Chemotherapy; Capecitabine; Gemcitabine; Cisplatin
Keywords: Cholangiocarcinoma; Adjuvant chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Active Comparator): Adjuvant Capecitabine
  Interventions: Drug: Capecitabine
- Gemcitabine plus cisplatin (Experimental): Adjuvant Gemcitabine plus Cisplatin
  Interventions: Drug: Gemcitabine plus cisplatin

INTERVENTIONS:
Drug: Gemcitabine plus cisplatin — Gemcitabine 1,000 mg/m2 and cisplatin 25 mg/m2 Day 1 and 8, every 3 weeks
  Other Names: Gemcitabine; Cisplatin
  Arms: Gemcitabine plus cisplatin
Drug: Capecitabine — Capecitabine 1,250 mg/m2 Day 1 to 14, every 3 weeks
  Arms: Capecitabine

SUMMARY:
There is no proven adjuvant treatment after curative surgical resection in patients with cholangiocarcinoma, although previous meta-analysis suggested potential survival benefit of adjuvant chemotherapy or radiotherapy in patients with lymph node-positive resected cholangiocarcinoma. Despite of lack of level 1 evidence and no data which regimen is optimal, adjuvant chemotherapy is widely used in daily practice setting. Based on this background, the investigators designed the randomized phase 2 trial comparing capecitabine and gemcitabine plus cisplatin in patients with resected lymph node-positive extrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years and older
* Histologically documented extrahepatic cholangiocarcinoma (perihilar or distal bile duct tumor)
* Microscopic or macroscopic surgical resection (ie., R0 or R1 resection)
* Regional lymph node metastasis according to the American Joint Committee on Cancer (AJCC) 7th edition
* No distant metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 1
* No prior chemotherapy or radiotherapy
* Serum CA 19-9 < 100 U/mL at the time of enrollment
* Adequate bone marrow function as defined by platelets ≥ 100 x 109/L and neutrophils ≥ 1.5 x 109/L
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal (ULN)
* Adequate hepatic function with serum total bilirubin < 2 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other non life-threatening cancer (i.e., prostate or thyroid cancer) except where treated with curative intent > 5 years previously without evidence of relapse Written informed consent to the study

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Histologies other than adenocarcinoma such as mixed hepatocellular carcinoma/cholangiocarcinoma, adenosquamous carcinoma or mixed adenocarcinoma/neuroendocrine carcinoma
* Intrahepatic cholangiocarcinoma or gallbladder cancer
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Female subjects who are pregnant or lactating, or males and females of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy from 2 weeks before receiving study drug until 3 months after receiving the last dose of study drug. A highly effective method of contraception is defined as having a low failure rate (< 1% per year) when used consistently and correctly.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
2-year disease-free survival | 2 years
  Proportion of patients without disease recurrence after 2 years

SECONDARY OUTCOMES:
Disease-free survival | 4 years
  Median time point that 50% of study patients recur
Toxicities (Adverse events related with chemotherapy) | 4 years
  Adverse events related with chemotherapy
Overall survival | 4 years
  Median time point that 50% of study patients is alive

CONTACTS AND LOCATIONS:
Overall Officials: Baek-Yeol Ryoo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horgan AM, Amir E, Walter T, Knox JJ. Adjuvant therapy in the treatment of biliary tract cancer: a systematic review and meta-analysis. J Clin Oncol. 2012 Jun 1;30(16):1934-40. doi: 10.1200/JCO.2011.40.5381. Epub 2012 Apr 23. PMID 22529261
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Ramirez-Merino N, Aix SP, Cortes-Funes H. Chemotherapy for cholangiocarcinoma: An update. World J Gastrointest Oncol. 2013 Jul 15;5(7):171-6. doi: 10.4251/wjgo.v5.i7.171. PMID 23919111
- [Background] Neoptolemos JP, Moore MJ, Cox TF, Valle JW, Palmer DH, McDonald AC, Carter R, Tebbutt NC, Dervenis C, Smith D, Glimelius B, Charnley RM, Lacaine F, Scarfe AG, Middleton MR, Anthoney A, Ghaneh P, Halloran CM, Lerch MM, Olah A, Rawcliffe CL, Verbeke CS, Campbell F, Buchler MW; European Study Group for Pancreatic Cancer. Effect of adjuvant chemotherapy with fluorouracil plus folinic acid or gemcitabine vs observation on survival in patients with resected periampullary adenocarcinoma: the ESPAC-3 periampullary cancer randomized trial. JAMA. 2012 Jul 11;308(2):147-56. doi: 10.1001/jama.2012.7352. PMID 22782416
- [Background] Patt YZ, Hassan MM, Aguayo A, Nooka AK, Lozano RD, Curley SA, Vauthey JN, Ellis LM, Schnirer II, Wolff RA, Charnsangavej C, Brown TD. Oral capecitabine for the treatment of hepatocellular carcinoma, cholangiocarcinoma, and gallbladder carcinoma. Cancer. 2004 Aug 1;101(3):578-86. doi: 10.1002/cncr.20368. PMID 15274071
- [Background] Petekkaya I, Gezgen G, Roach EC, Solak M, Gullu I. Long-term advanced cholangiocarcinoma survivor with single-agent capecitabine. J BUON. 2012 Oct-Dec;17(4):796. No abstract available. PMID 23335544
- [Derived] Jeong H, Oh JH, Ahn HS, Ryoo BY, Kim KP, Jeong JH, Park I, Hwang DW, Lee JH, Song KB, Lee W, Kim KH, Moon DB, Song GW, Jung DH, Hong SM, Park CW, Baek IP, Cho YS, Kim K, Sung CO, Yoo C. Proteogenomic profiling predicts outcomes of adjuvant chemotherapy in extrahepatic cholangiocarcinoma. J Hepatol. 2026 Jan;84(1):122-134. doi: 10.1016/j.jhep.2025.07.031. Epub 2025 Aug 11. PMID 40803577
- [Derived] Yoo C, Jeong H, Jeong JH, Kim KP, Lee S, Ryoo BY, Hwang DW, Lee JH, Moon DB, Kim KH, Lee SS, Song TJ, Oh D, Lee MA, Chon HJ, Lee JS, Laliotis G, Rivero-Hinojosa S, Spickard E, Renner D, Dutta P, Palsuledesai CC, Sharma S, Malhotra M, Jurdi A, Liu MC. Circulating tumor DNA status and dynamics predict recurrence in patients with resected extrahepatic cholangiocarcinoma. J Hepatol. 2025 May;82(5):861-870. doi: 10.1016/j.jhep.2024.10.043. Epub 2024 Nov 10. PMID 39532185